CLINICAL TRIAL: NCT04920838
Title: Early Treatment of Vulnerable Individuals With Non-Severe SARS-CoV-2 Infection: A Multi-Arm Multi-Stage Randomized Trial (MAMS) to Evaluate the Effectiveness of Several Specific Treatments in Reducing the Risk of Clinical Worsening or Death in Sub-Saharan Africa (COVERAGE-Africa)
Brief Title: Early Treatment of Vulnerable Individuals With Non-Severe SARS-CoV-2 Infection
Acronym: COVERAGE-A
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University of Bordeaux (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); PACCI Program (Other); Alliance for International Medical Action (Other); Centre Muraz (Other); Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS COV33 COVERAGE-Africa
Record Dates: First submitted 2021-05-04; First posted 2021-06-10 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Covid19 Drug Treatment; Severe Acute Respiratory Syndrome Coronavirus 2; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide; Telmisartan; Tablets; Acetaminophen; Fluoxetine

STUDY DESIGN:
Intervention Model Description: This is a multicentre, multiple country, randomised, open-label, adaptive, platform clinical study aiming to determine the efficacy and safety of various treatment regimens for prevention of the need for hospitalisation for specialised care due to severe progression of COVID-19.
  The study is designed with the ability to incorporate the adding or dropping of treatment arms and that will include similar inclusion and non-inclusion criteria, the same primary and secondary endpoints, common data entry procedures, a shared database and a single statistical methodology for analysis of the primary endpoint.
Masking Description: Investigators and all the staff in clinical sites will not be masked. Data manager and statician will not be masked too. However, the sponsor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Paracetamol (Active Comparator): Patients in this arm will receive paracetamol during 14 days
  Interventions: Drug: Paracetamol
- Nitazoxanide and Ciclésonide (Experimental): Patients in this arm will receive the combination of ciclezonide (Alvesco® 160 µg ) / nitazoxanide (Netazox® 500 mg) during 14 days
  Interventions: Drug: Nitazoxanide and Ciclésonide
- Telmisartan (Experimental): Patients in this arm will receive telmisartan (Micardis® 20 mg) during 10 days
  Interventions: Drug: Telmisartan 20Mg Oral Tablet
- Fluoxétine and Budésonide (Experimental): Patients in this arm will receive the combination of Fluoxétine (Fluoxétine Arrow® 40 mg ) / Budésonide (Budecort® 2*400 mcg) during 7 days
  Interventions: Drug: Fluoxétine and Budésonide

INTERVENTIONS:
Drug: Nitazoxanide and Ciclésonide — Inhaled Ciclésonide: 320 mcg BID per day and Oral Nitazoxanide:2000 mg tablets daily (divided into two daily intakes of two tablets of nitazoxanide 500 mg) during 14 days.
  Arms: Nitazoxanide and Ciclésonide
Drug: Telmisartan 20Mg Oral Tablet — 20 mg tablet daily
  Arms: Telmisartan
Drug: Paracetamol — Tablets containing 500 mg of paracetamol. One to two tablets every 4-6 hours as required, to a maximum of 6 tablets (3 grams) daily in divided doses.
  Duration of treatment: up to 14 days
  Arms: Paracetamol
Drug: Fluoxétine and Budésonide — Inhaled Budésonide: 400mcg BID per day and oral Fluoxétine : 80mg tablets daily (divided into two daily intakes of two tablets of Fluoxétine 40 mg) during 7 days.
  Arms: Fluoxétine and Budésonide

SUMMARY:
Coverage Africa is a nested study in the large Anticov platform trial that aims to generate data on new early treatment strategies for mild/moderate COVID-19 patients in resource-limited-settings to reduce the number progressing to severe forms requiring hospitalization, thereby relieving the burden on health care systems and contributing to "flattening the curve" in contexts where none pharmaceutical intervention such as quarantine are difficult to implement in large urban settings. Treating early when the virus is still present might also limit transmission. Coverage Africa will be conducted in Guinea and Burkina Faso.

The main objective is to conduct an open-label, multicenter, randomized, adaptive platform trial to test the safety and efficacy of several marketed products, including antiviral therapies versus control in mild/moderate of coronavirus disease 2019 (Covid-19) in resource-limited-settings.

The study aims to recruit 600 patients in both countries, one site in Guinea and two sites in Burkina Faso.

The current assessed treatments are now the association of Fluoxétine/Budésonide compared with a control arm: paracetamol.

The adaptive design trial will allow for the removal of drugs, or the addition of new study arms when new data becomes available. Data on the primary efficacy parameters and safety will be integrated with the primary endpoint based on an oxygen saturation percentage (SpO2) ≤ 93% or death within 14 days after randomization to treatment, including death for any reason.

Study will run until August 2022. However, with the proposed adaptive design, the study could also be interrupted for success earlier than planned with the identification of a treatment that significantly reduces hospitalization rate as evidence by results from the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age at the time of screening or >= 40 years and presenting at least one comorbidity : high blood pressure; a known obesity and/ or a known and treated diabete.
* SARS-CoV-2 infection confirmed by molecular biology (RT-PCR on a nasopharyngeal or oropharyngeal swab) or by antigen test validated in the country according to national guidelines
* A viral syndrome with or without uncomplicated pneumonia, defined as blood oxygen saturation level (SpO2) >=94%.
* Mild Covid-19 symptoms with an onset < 7 days before inclusion.
* Signed written consent from the patient or his/her representative.
* No need an oxygen therapy according to international guidelines (WHO Progression Scale, grade 2 to 4)
* Accepting and having the ability to be reached by telephone throughout the study.
* Having designated a contact person who can be contacted in case of emergency.
* Accepted to be reached by phone along throughout the study

Exclusion Criteria:

* Blood oxygen saturation level (SpO2) < 94%.
* Known hypersensitivity to investigational products
* Chronic treatment with inhaled corticosteroids (up to 30 days)
* Known history of renal or hepatic failure
* Abnormal physical examination findings:

  * respiratory rate < 25 per minute;
  * Clinical hypotension with associated signs justifying hospital care
* Feeling unwell for more than 7 days prior to screening.
* End-organ compromise requiring admission to a resuscitation or continuous care unit or short-term life-threatening comorbidity with life expectancy < 3 months.
* For any new antiviral included in the study, prior treatment with the antiviral, presence of contraindication to its use or intake of concomitant medication proscribed with its use.
* Patients with known suicidal thoughts, severe psychiatric disorders or major depression that is uncontrolled or controlled by one of the prohibited drugs
* Known history of long QT syndrome or severe ventricular cardiac arrhythmia (ventricular tachycardia, patients with recovered ventricular fibrillation)
* Unwilling or unable to comply with the requirements of the study protocol at any time during the study, e.g. no access to or not comfortable with use of a smartphone or with answering questions using a telephone, in the opinion of the Investigator or cannot use an inhalation chamber.
* Any other reason that makes it impossible to monitor the patient during the study.
* Enrolled in other clinical trials with unregistered drugs or with registered drugs that may interact with any of the study IPs or are contraindicated as concomitant therapy within the last 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
SpO2 ≤ 93% within 14 days | From inclusion (day 0) to day 14.
  Percentage of participant presenting an oxygen saturation percentage (SpO2) ≤ 93% or death within 14 days after randomization to treatment.
Death within 14 days | From inclusion (day 0) to day 14.
  Percentage of participant dead within 14 days after randomization to treatment, including death for any reason.

SECONDARY OUTCOMES:
Death within 28 days | From inclusion (day 0) to day 28.
  Percentage of participant dead within 28 days after randomization to treatment, including death for any reason.
Occurence of at least one grade 3 or 4 clinical or biological adverse event within 14 days | From inclusion (day 0) to day 14.
  Occurence of at least one grade 3 or 4 clinical or biological adverse event within 14 days
Number of hospitalizations due to severe progression | From inclusion (day 0) to day 28.
  Hospitalisation due to aggravation of COVID-19, including hospitalisation's reason as described below
  * Request of mechanical ventilation and/or Intensive Care Unit (ICU)
  * Non-ICU hospitalisation, requiring supplemental oxygen
  * Non-ICU hospitalisation, not requiring supplemental oxygen

CONTACTS AND LOCATIONS:
Locations (2):
- Centre Muraz/INSP, Bobo-Dioulasso, Burkina Faso
- Centre de traitement des maladies à tendance épidémique de Gbessia, Conakry, Guinea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Doucet MH, Songbono CT, Plazy M, Martin C, Fritzell C, Sow MS, Traore FA, Jaspard M, Poda A, Malvy D, Marcy O, Delamou A, Orne-Gliemann J. Perceptions of COVID-19 among communities of Conakry (Guinea): a qualitative study exploring the context of the ANRS COV33 Coverage-Africa therapeutic trial. BMJ Open. 2022 Dec 27;12(12):e061715. doi: 10.1136/bmjopen-2022-061715. PMID 36574985